CLINICAL TRIAL: NCT01003600
Title: Colorectal Cancer Survivors' Needs and Preferences for Survivorship Information
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Queens Cancer Center of Queens Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 09-133
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Survivorship; Quality of Life; Questionnaire; 09-133
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Questionnaire: This study is a cross-sectional survey study to be administered to adults who completed treatment for nonmetastatic colorectal cancer at MSKCC or at Queens Cancer Center (QCC) at Queens Hospital between 6 months and 2 years ago and have no evidence of disease at the time of study enrollment.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — The questionnaire will be administered by telephone and will take approximately 20-30 minutes. The questionnaire will elicit survivor responses along five domains: knowledge about diagnosis and treatment, knowledge about ongoing risks and recommended testing, history of health care utilization since the end of treatment, preferences for relevant information about these topics, and employment after the end of cancer treatment.
  Other Names: The questionnaire will be administered using a Computer Assisted Telephone Interview (CATI); system. The CATI form of the questionnaire enables the interviewer to read aloud from a script and; enter responses into the computer in real-time, regardless of whether the interview is conducted on the; phone or in person. The CATI form of the questionnaire enables the interviewer to read aloud from a; script and enter responses into the computer in real-time, regardless of whether the interview is; conducted on the phone or in person.

SUMMARY:
We are doing this study to learn more about colon and rectal cancer survivors. We want to know if survivors want more information about life after cancer. Do cancer survivors want to know more about their own cancer? Do cancer survivors want to know about their treatment? Do cancer survivors want to know what health care they should get in the future? We want to know what information to give to cancer survivors when they finish treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at diagnosis
* Diagnosed with first primary colorectal cancer (stage I-III)
* Completed last treatment for colorectal cancer (surgery, chemotherapy, or radiation) at least 6 months and no more than 2 years before the date of study enrollment
* Able to speak English, because questionnaire is only available in English
* Able to provide informed consent
* Received all treatment for colorectal cancer at MSKCC or QCC or, surgical treatment at an outside facility, and all other treatment (chemotherapy or radiation) at MSKCC or QCC

Exclusion Criteria:

* Undergoing active treatment for colorectal cancer
* Diagnosed with metastatic colorectal cancer
* Prior history of colorectal or any other cancer (except non-melanoma skin cancer)
* Diagnosed with new or recurrent colorectal or other cancer after the primary colorectal cancer diagnosis
* Received a survivorship care plan from the treating institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who completed treatment for nonmetastatic colorectal cancer at MSKCC or at Queens Cancer Center (QCC) at Queens Hospital
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2009-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Assess colorectal cancer survivors' basic knowledge of their own cancer history, including date of diagnosis, stage, and treatments received. | 6 months to 2 years after completion of treatment

SECONDARY OUTCOMES:
Assess survivors' knowledge of medical issues relevant to colorectal cancer survivors. | 6 months to 2 years after completion of treatment
Describe the types of health care providers that survivors have visited since completing treatment for colorectal cancer. | 6 months to 2 years after completion of treatment
Assess survivors' preferences for the content, format, and delivery of survivorship care plans. | 6 months to 2 years after completion of treatment
Assess whether survivors who had concerns about working after cancer treatment spoke with health care professionals about their concerns. | 6 months to 2 years after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Talya Salz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm